CLINICAL TRIAL: NCT00098111
Title: A Double-Blinded, Randomized, Parallel Arm, Dose Ranging Study of IMURAN in Subjects With Active Crohn's Disease Requiring Treatment With Prednisone: A Crohn's Disease Optimal Range Dose of IMURAN Study (ACORDIS)
Brief Title: Imuran (Azathioprine) Dose-Ranging Study in Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Bruce Sands, Associate Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: FD-R-02555-01; Grant # 2555
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; inflammatory bowel disease; IMURAN; azathioprine
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Azathioprine 0.5 mg/kg body weight (Active Comparator)
  Interventions: Drug: azathioprine
- Azathioprine 2.5 mg/kg body weight (Active Comparator)
  Interventions: Drug: azathioprine
- Azathioprine 3.5 mg/kg body weight (Active Comparator)
  Interventions: Drug: azathioprine

INTERVENTIONS:
Drug: azathioprine

SUMMARY:
The purpose of this study is to identify an optimal weight based dose of azathioprine that is safe and effective in the treatment of subjects with active Crohn's disease requiring treatment with corticosteroids, and for maintaining remission in those subjects.

DETAILED DESCRIPTION:
DESCRIPTION: Medical therapy for Crohn's disease is of variable success in ameliorating the cardinal symptoms of the disease (diarrhea, abdominal pain), in treating extraintestinal manifestations (fatigue, anorexia, fever, weight loss, arthralgias, skin, eye, liver and kidney manifestations), and in preventing complications (stricture, fistula, abscess). Currently, therapy is most often implemented in a stepwise fashion, progressing through anti-inflammatory medications (sulfasalazine, mesalamine), antibiotics (metronidazole, ciprofloxacin), corticosteroids, immunomodulatory or immunosuppressive medications, including thioguanine compounds (6 mercaptopurine or its prodrug azathioprine), methotrexate, and finally, infliximab (anti-tumor necrosis factor). A common approach is the gradual addition of more potent medications to agents that are believed to be safer, but may also be less effective. Despite the current approach to medical therapy in Crohn's disease, a substantial number of patients-from 20 to 40%-require surgery within 3 years of diagnosis, excluding those requiring surgery at the time of diagnosis. Nearly 80% of patients require surgery by 20 years from the onset of disease.

Corticosteroids have long been a mainstay of therapy in Crohn's disease although side effects are frequently observed with both short term and long-term use. Potential side effects are well-described, and may include relatively minor problems such as insomnia and acne, as well as more serious adverse effects, including hypertension, narrow-angle glaucoma, depression, weight gain, adrenal suppression, Cushing's syndrome, diminished bone mineral density, and infections.

Azathioprine is often used to treat patients with steroid resistant or dependent Crohn's disease. Azathioprine is used as a steroid sparing agent, as treatment for active, inflammatory disease, for maintenance of remission, as therapy for perforating disease (fistulae), and for specific extraintestinal manifestations. To date, however, randomized, controlled clinical studies assessing a range of doses of azathioprine in Crohn's disease have not been conducted. The optimal weight-based dose is not known.

EXPECTED CONTRIBUTION: This study will identify an optimal weight based dose of azathioprine for treatment of patients with active Crohn's disease requiring treatment with corticosteroids.

STUDY HYPOTHESIS: An optimal weight-based dose of azathioprine will induce and maintain remission in subjects with steroid-dependent Crohn's disease.

COMPARISON: Three different doses of azathioprine will be compared in this study (0.5, 2.5, and 3.5mg/kg/day). Subjects will take the study medication for 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 14 years old, including women of childbearing potential who are not pregnant or nursing at the time of enrollment.
* Body weight between 40 and 100 kg (88-220 lbs), inclusive.
* Subjects diagnosed with Crohn's disease, based upon the criteria of Lennard-Jones, for at least a 3-month period. The date of diagnosis will be the date of the first diagnostic test that confirms the diagnosis of Crohn's disease. Subjects with a diagnosis of less than 3 months may be considered after review of primary diagnostic data by the study safety monitor.
* Need for treatment with oral prednisone, based upon the treating physician's clinical judgment, for active Crohn's disease as indicated by a (Crohn's Disease Activity Index) CDAI between 200 and 450, inclusive; OR Currently being treated with prednisone for at least 4 weeks with a stable dose of 40mg/day or less for at least 2 weeks, or budesonide (Entocort EC) 9 mg/day for at least 4 weeks with a stable dose for at least 4 weeks, and active Crohn's disease as indicated by a CDAI between 200 and 450, inclusive.
* Able to swallow tablets.
* Able to provide written informed consent (subjects ≥ 18 years old) or in the case of a minor provide parental consent along with child assent (subjects 14-17 years old).
* If sexually active, willing to comply with effective contraception during the study; or is abstinent.

Exclusion Criteria:

* Diagnosis of indeterminate, microscopic, lymphocytic, collagenous, or ulcerative colitis.
* Previous or current therapy with 6-mercaptopurine, azathioprine, thioguanine, methotrexate, cyclosporine, tacrolimus, thalidomide or mycophenolate mofetil.
* Previous or current treatment with infliximab.
* Treatment with narcotic pain medications. (Anti-diarrheal agents such as loperamide and diphenoxylate are permitted, providing that the dose is not increased while on protocol.)
* Subjects with short gut syndrome (defined as requiring oral or parenteral supplemental or total nutrition in order to maintain stable body weight, or more than 100 cm of small bowel resected).
* Subjects with obstructive symptoms or demonstrated stenosis and prestenotic dilatation on barium study.
* Subjects with active infection.
* Subjects with a stoma.
* Subjects with heterozygous or recessive homozygous genotype for TPMT.
* Poor access for peripheral venous phlebotomy.
* History of pancreatitis, except for self-limited episodes from a known cause, such as gallstone pancreatitis.
* White blood cell count (WBC) <4.5 x 10^9/L, hemoglobin <8 gm/dL, Platelets (PLT) <100,000/mm3 at screening (or within the previous 6 months, if known).
* History of abnormal liver function tests, including aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times upper limit of normal, alkaline phosphatase >2 times upper limit of normal, total bilirubin >2.5 mg/dL at screening (or within the previous 6 months, if known).
* Subjects needing treatment with orally administered corticosteroids for the treatment of other medical conditions. Inhaled or dermatologic preparations are acceptable.
* History of HIV infection (if known) or opportunistic infection.
* History of cancer, with the exception of basal cell carcinoma of the skin.
* Concurrent treatment, or need for treatment, with allopurinol.
* Women who are pregnant or nursing at the time of eligibility screening, or who intend to be during the study period.
* Inability to comply with planned schedule of study visits.
* Participation in a clinical trial within the past 6 months.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To identify an optimal weight-based dose of azathioprine for the treatment of active Crohn's disease and for maintaining remission in those subjects.

SECONDARY OUTCOMES:
To characterize prospectively the predictive value of erythrocyte thioguanine nucleotide levels for response to azathioprine in who are wild type for the (thiopurine methyltransferase) TPMT gene
To explore the relationship of 6-thioguanine (TGN) levels to TPMT enzyme activity
To determine the effect of azathioprine dose upon time to relapse among subjects in remission induced by a course of prednisone
To prospectively determine the rate of adverse events associated with a range of doses of azathioprine
To preliminarily identify genetic polymorphisms associated with therapeutic response or toxicity to azathioprine.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce E Sands, M.D.,M.S., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States